CLINICAL TRIAL: NCT05663333
Title: Histopathological Analysis of Temporal Artery Biopsy Following Dynamic Full-field Optical Coherence Tomography, a Comparison to Conventional Histopathological Findings in Patients With Suspected Giant Cell Arteritis
Brief Title: Histopathological Analysis of Temporal Artery Biopsy Following Dynamic Full-field Optical Coherence Tomography, a Comparison to Conventional Histopathological Findings in Patients With Suspected Giant Cell Arteritis (DOCTA)
Acronym: DOCTA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier William Morey - Chalon sur Saône (Other)
Collaborators: Centre Hospitalier de Mâcon (Other)
Responsible Party: Principal Investigator, Thomas Maldiney, Doctor, Centre Hospitalier William Morey - Chalon sur Saône
Other Study IDs: DOCTA
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Giant Cell Arteritis; Tomography, Optical Coherence
Keywords: Giant Cell Arteritis; Temporal Artery Biopsy; Full-field Optical Coherence Tomography
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DOCTA cohort: Patients > 50 years of age with suspected giant cell arteritis requiring temporal artery biopsy in the dermatology department
  Interventions: Other: Dynamic full-field optical coherence tomography analysis of temporal artery biopsy

INTERVENTIONS:
Other: Dynamic full-field optical coherence tomography analysis of temporal artery biopsy — Dynamic full-field optical coherence tomography analysis of temporal artery biopsy in the dermatology department before conventional histopathological analysis

SUMMARY:
Giant cell arteritis (GCA) is a type of large vessel granulomatous vasculitis responsible for the inflammation of the aorta and the branches of the external carotid, notably temporal arteries. The diagnosis of GCA relies upon the identification of vasculitis following histopathological analysis of temporal artery biopsy (TAB) showing mononuclear cells infiltration, fragmentation of the internal elastic lamina as well as significant intimal hyperplasia. Apart from its lack of sensitivity, one of the weaknesses of TAB is the delay in obtaining the result due to the time required to prepare the sample for histological analysis. Pursuing the idea to improve TAB performances, our group recently demonstrated the use of full-field optical coherence tomography (FF-OCT) to visualize structural changes associated with the inflammatory processes of GCA. The present work suggests a further use of dynamic FF-OCT on TAB for a direct visualization of the mononuclear cells infiltration to ensure rapid on-site diagnosis of GCA.

ELIGIBILITY:
Inclusion Criteria:

* patient > 50 years of age with suspected giant cell arteritis who received temporal artery biopsy between start study date and primary completion date

Exclusion Criteria:

* inability to perform dynamic full-field optical coherence tomography observation at the moment of temporal artery biopsy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient > 50 years of age with suspected giant cell arteritis who received temporal artery biopsy
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Histopathological analysis of healthy temporal artery biopsy with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following temporal artery biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify the normal structures of a temporal artery biopsy, i.e. the tripartite architecture with a clear distinction between intima (endothelial cells), media (vascular smooth muscle cells) and adventitia, both internal and external elastic lamina, and vasa vasorum

SECONDARY OUTCOMES:
Histopathological features of giant cell arteritis with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following temporal artery biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify histopathological features of giant cell arteritis, i.e. infiltration of mononuclear cells in the three layers of the artery, fragmentation of the internal elastic lamina, intimal hyperplasia and neoangiogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldiney, Principal Investigator — Centre Hospitalier William Morey - Chalon sur Saône
Locations (1):
- Centre Hospitalier William Morey - Chalon sur Saône, Chalon-sur-Saône, Saône-et-Loire, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maz M, Chung SA, Abril A, Langford CA, Gorelik M, Guyatt G, Archer AM, Conn DL, Full KA, Grayson PC, Ibarra MF, Imundo LF, Kim S, Merkel PA, Rhee RL, Seo P, Stone JH, Sule S, Sundel RP, Vitobaldi OI, Warner A, Byram K, Dua AB, Husainat N, James KE, Kalot MA, Lin YC, Springer JM, Turgunbaev M, Villa-Forte A, Turner AS, Mustafa RA. 2021 American College of Rheumatology/Vasculitis Foundation Guideline for the Management of Giant Cell Arteritis and Takayasu Arteritis. Arthritis Rheumatol. 2021 Aug;73(8):1349-1365. doi: 10.1002/art.41774. Epub 2021 Jul 8. PMID 34235884
- [Background] Maldiney T, Greigert H, Martin L, Benoit E, Creuzot-Garcher C, Gabrielle PH, Chassot JM, Boccara C, Balvay D, Tavitian B, Clement O, Audia S, Bonnotte B, Samson M. Full-field optical coherence tomography for the diagnosis of giant cell arteritis. PLoS One. 2020 Aug 31;15(8):e0234165. doi: 10.1371/journal.pone.0234165. eCollection 2020. PMID 32866179